CLINICAL TRIAL: NCT03370263
Title: BENLYSTA for Intravenous Injection / Subcutaneous Injection Special Drug Use Investigation
Brief Title: BENLYSTA® Special Drug Use Investigation
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 207735
Record Dates: First submitted 2017-12-06; First posted 2017-12-12 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Benlysta, systemic lupus erythematosus, safety, efficacy
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — belimumab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Benlysta intravenous (IV): This arm will include subjects who will receive Benlysta IV. Observation period per subject will be for 52 weeks from start of Benlysta administration.
  Interventions: Drug: Benlysta
- Benlysta subcutaneous (SC): This arm will include subjects who will receive BENLYSTA SC. Observation period per subject will be for 52 weeks from start of Benlysta administration.
  Interventions: Drug: Benlysta

INTERVENTIONS:
Drug: Benlysta — Benlysta will be administered intravenously or subcutaneously.

SUMMARY:
The objective of this study is to collect and assess the information about long-term safety and effectiveness of Benlysta for intravenous injection and Benlysta for subcutaneous injection (hereinafter referred to as "Benlysta") in daily clinical practice. The aim of conducting this drug use investigation (DUI) in all subjects until data are accumulated from a certain number of subjects after Benlysta being marketed, data will be collected on safety and effectiveness of Benlysta in an early stage and thereby to take the necessary measures for proper use of Benlysta. Approximately 600 subjects will be enrolled in to this study. The observation period per subject will be 52 weeks from the start of Benlysta administration. BENLYSTA is the registered trademark of GlaxoSmithKline (GSK) group of companies.

ELIGIBILITY:
Inclusion Criteria:

* The study will include all subjects to whom Benlysta is administered. In addition, among subjects who start administration after launch, those to whom Benlysta has already administered before the conclusion of the contract and those who has already started administration at diagnosis, because of hospital transfer, etc. will be included as well.

Exclusion Criteria:

* N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will include all subjects to whom Benlysta is administered. In addition, among subjects who start administration after launch, those to whom Benlysta has already administered before the conclusion of the contract and those who has already started administration at diagnosis, because of hospital transfer, etc. will be included as well.
Sampling Method: Probability Sample
Enrollment: 1514 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2025-09-26 (Actual); Study Completion 2025-09-26 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Safety of Estrogens in Lupus Erythematosus National Assessment Systemic Lupus Erythematosus Disease Activity Index (SELENA SLEDAI) | Baseline and up to 52 weeks
  The Systemic Lupus Erythematosus Disease Activity Index (SLEDAI) is a validated index for assessing Systemic Lupus Erythematosus (SLE) disease activity. It is a weighted index in which signs and symptoms, laboratory tests, and physician's assessment for each of 9 organ systems are given a weighted score and summed, if present at the time of the visit or in the preceding 10 days. Modified version of SLEDAI is Safety of Estrogen in Lupus National Assessment (SELENA) SLEDAI where the maximum theoretical score for the SELENA SLEDAI was 105 with 0 indicating inactive disease.
Change from Baseline in Physician's Global Assessment (PGA) score | Baseline and up to 52 weeks
  The PGA is a 0 to 30 centimeters (cm) visual analogue scale (VAS). The investigator will assess the subject's global disease activity, and draw a vertical line between 0 (none) and 3 (severe) where 0 is none (no disease activity), 1 is mild, 2 is moderate and 3 is severe (worst lupus disease imaginable).
Change from Baseline in Lupus Impact Tracker score | Baseline and up to 52 weeks
  The investigator will interview subjects about their conditions in the previous one month using Lupus Impact Tracker, the impact on daily living will be assessed using a 5-point scale of 0 (none of the time) to 4 (all of the time).
Number of subjects with abnormal change in laboratory parameters | Baseline and up to 52 weeks
  Information will be collected for number of subjects with abnormal changes in laboratory parameters.
Number of subjects with adverse events (AE) and serious adverse events (SAE) | Up to 52 weeks
  AE is any untoward medical occurrence in a subject or clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is any untoward medical occurrence that, at any dose results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect or is medically significant.
Number of subjects with adverse drug reactions (ADR) of events defined as a priority study matter | Up to 52 weeks
  An adverse drug reaction (ADR) is an unwanted or harmful reaction experienced following the administration of a drug or combination of drugs under normal conditions of use and is suspected to be related to the drug. Following will be considered as priority study matter: Serious hypersensitivity, Serious infections (including tuberculosis [TB], pneumonia, pneumocystis pneumonia [PCP], sepsis, and opportunistic infection [OI]), Reactivation of hepatitis B (HB) virus, Progressive multifocal leukoencephalopathy (PML), Interstitial pneumonitis (IP), Malignant tumor (MT), Depression and events related to suicide/self-injury.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Hiroshima, Japan

IPD SHARING:
Plan to Share IPD: No